ID: COPD-141316051 NCT02251496

**COPD: Oral Nutrition Supplements vs. Energy- and Protein Dense in Between Meal Snacks.** 

## Statistical analysis

All statistical analyses were undertaken using IBM SPSS Statistics 24 and the level of significance was set at 0.05. Our original power calculations were based on the primary outcome of difference in weight gain between the groups and change in weight to one year. Due to low recruitment rate and lower participation rates than expected, post-hoc power calculations were performed based on our results. The Kolmogorov-Smirnov test was used to test data normality. The independent t-test was used to test for differences between continuous data at baseline and the Pearson's chi-squared test was used for categorical data. Intention-to-treat analyses were conducted where the last observations were carried forward and used to assess treatment efficacy. All patients with at least two measures (baseline and one other) were included. Repeated measures ANCOVA was conducted to analyse mean changes in each follow up.